CLINICAL TRIAL: NCT03122197
Title: A Phase 0/1 Pharmacokinetic and Pharmacodynamics and Safety and Tolerability Study of Letrozole in Combination With Standard Therapy in Recurrent High Grade Gliomas
Brief Title: Study of Letrozole in Recurrent Gliomas
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Trisha Wise-Draper, Principal Investigator, University of Cincinnati
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCCI-BN-16-01
Record Dates: First submitted 2017-04-10; First posted 2017-04-20 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms | interventions — Letrozole; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Letrozole (Experimental): The BN-16-01 main study treatment starting dose will be 2.5mg administered orally once daily. Daily doses up to 10mg and single doses of 30mg have been shown to be safe in prior studies and therefore we expect that letrozole doses up to 20mg in this study will be safe.
  The recommended phase II dose (RP2D) will be considered the dose that results in ≥ 2uM letrozole concentration in the tumor or the highest dose achieved (20mg daily for cohort level 7) with < 2/6 patients with DLTs. This dose will be planned for future phase II studies to determine potential efficacy.
  Interventions: Drug: Letrozole Oral Tablet
- Letrozole and temozolomide (Experimental): Phase 1 expansion cohort of letrozole 15mg administered in combination with 50 mg/m2 metronomic temozolomide (TMZ) in patients with high grade gliomas. Letrozole 15mg will be administered orally once daily for a 7-day lead-in period. After 7 days subjects will continue letrozole in combination 50 mg/m2 TMZ administered orally once daily.
  Interventions: Drug: Letrozole Oral Tablet; Drug: Temozolomide
- Previously Received letrozole and temozolomide (Experimental): Phase 1 expansion cohort of two identified subjects with gliomas who previously participated in the main study UCCI-BN-16-01 who received as physician's choice of treatment 50 mg/m2 TMZ in combination with dosing of 15 mg letrozole.
  Interventions: Drug: Letrozole Oral Tablet; Drug: Temozolomide

INTERVENTIONS:
Drug: Letrozole Oral Tablet — Administration: Letrozole will be given orally once daily.
  Other Names: Femara
Drug: Temozolomide — 50 mg/m2 TMZ administered orally once daily
  Other Names: Temodar
  Arms: Letrozole and temozolomide; Previously Received letrozole and temozolomide

SUMMARY:
The purpose of this study is to determine the ability of letrozole to penetrate the blood brain barrier and concentrate in gliomas.

DETAILED DESCRIPTION:
Nine to forty-two (42 patients only if every cohort required expansion) total patients were planned for the main BN-16-01 phase 0/1 study to explore the ability of letrozole to penetrate the blood brain barrier and gliomas. As of November 2023 The BN-16-01 main study has completed active recruitment (20 subjects were accrued) and all safety and pharmacokinetics data have been analyzed with subsequent publications pending. Characterization of the safety and pharmacokinetics of letrozole in combination with standard of care treatments, such as TMZ has been completed for the main study and provides the rationale for initiation of a sub-study.

A new sub-study "Letrozole and Temozolomide" expansion cohort has been opened to accrual. This Phase 1 expansion cohort of letrozole 15mg administered in combination with 50 mg/m2 metronomic temozolomide (TMZ) in patients with high grade gliomas. 19 subjects total (2 historical subjects from the main study and 17 new accruals) will be enrolled into this expansion cohort.

ELIGIBILITY:
Inclusion Criteria

1. Radiographically, histologically or cytologically confirmed recurrent brain high grade glioma with plan for resection or biopsy.

   - Inclusion #1 for Sub-study Only: Radiographically, histologically or cytologically confirmed recurrent brain high grade glioma.
2. Age >18 years.
3. ECOG performance status 0 -2 (Karnofsky >60%, see Appendix A).
4. CBC/differential obtained within 28 days prior to registration on study, with adequate bone marrow function defined as follows:

   * Absolute neutrophil count (ANC) ≥ 1,000 cells/mm3;
   * Platelets ≥ 100,000 cells/mm3;
   * Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable).
5. Adequate hepatic function, defined as follows:

   * Total bilirubin < 2 x institutional ULN within 14 days prior to registration;
   * AST or ALT < 3 x institutional ULN within 14 days prior to registration.
6. Adequate renal function, defined as GFR > 30 ml/min or Cr < 1.5.
7. Negative serum pregnancy test within 2 weeks prior to registration for women of childbearing potential.
8. Imaging prior to treatment including MRI of brain (with contrast preferred but not required).
9. Ability to understand and the willingness to sign a written informed consent document.
10. Inclusion #10 for Sub-study Only: Measurable disease per RANO criteria within 28 days of starting treatment on this study.

Exclusion Criteria

1. Patients may not be receiving any other investigational agents.
2. History of allergic reactions attributed to letrozole or other agents used in study.

   Exclusion #2 for Sub-study Only: History of allergic reactions attributed to letrozole or TMZ.
3. Uncontrolled intercurrent illness including, but not limited to, ongoing significant or serious active cardiovascular disease (CHF exacerbation, unstable angina or MI in last 6 months), or infection including the diagnosis of AIDS or active hepatitis B or C infection, or psychiatric illness or medical or personal conditions that in the opinion of the investigator would limit the patient's ability to participate.
4. Patients attempting to conceive, and pregnant or nursing women are excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2017-05-16 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Overall Letrozole AUC in tumor tissue. | 5 days
  Pharmacokinetic modeling will be used to determine the overall AUC in the tumor tissue to assess for letrozole penetration through blood brain barrier.
Progression free survival in letrozole and temozolomide combination | 6 months
  Sub-study expansion cohort only: Progression free survival using RANO criteria at 6 months from the start of the combination of 15 mg letrozole and 50 mg/m2 temozolomide.

SECONDARY OUTCOMES:
Adverse Events | The time patients remain on treatment until 30 days after treatment completed
  The number of patients with treatment related toxicity will be assessed using CTCAE v4.0
Progression free Survival | From start of treatment until time of progression assessed up to 1 year
  Patients will be followed for response using RANO criteria to determine time from start of treatment to progression.
Overall Survival | From start of treatment until time of death assessed up to 1 year
  Patients will be followed from start of treatment until time of death

CONTACTS AND LOCATIONS:
Overall Officials: Trisha Wise-Draper, MD, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No